CLINICAL TRIAL: NCT03629002
Title: BIOLOGICAL EXPLORATION OF THE VASCULAR FRACTION FROM THE ADIPOSE TISSUE OF PATIENTS WITH SCLERODERMIA IN THE CONTEXT OF THE DEVELOPMENT OF AN INNOVATIVE CELLULAR THERAPY FOR THE TREATMENT OF FUNCTIONAL HANDICAP OF THE HAND
Brief Title: BIOLOGICAL EXPLORATION OF THE VASCULAR FRACTION FROM THE ADIPOSE TISSUE OF PATIENTS WITH SCLERODERMIA
Acronym: sclerabio
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-06; IDRCB (Other: 2018-A00150-55)
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Systemic Scleroderma
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stromal vascular fraction obtained from adipose tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with systemic scleroderma: Use of the biological collection of the vascualire stromal fraction of the SCLERADEC 2 clinical trial.
  Interventions: Biological: Study of the gene expression profile
- healthy volunteers: Recovery of a sample of adipose tissue during a liposuction operation in a context of routine cosmetic surgery.
  Interventions: Biological: Study of the gene expression profile

INTERVENTIONS:
Biological: Study of the gene expression profile — qPCR analysis

SUMMARY:
The overall objective is to propose a comprehensive analysis of the biological properties of the stromal vascular fraction evaluated in the SCLERADEC 2 clinical trial (n = 15 available) and preserved in the biological collection, compared to healthy donors (n = 10). This characterization will focus on the exploration of the phenotypic and functional characteristics of the main cellular subpopulations present in the stromal vascular fraction of scleroderma patients likely to be associated with a better regenerative vascular or anti-fibrotic activity of the cell therapy product.

The main objective will be to validate whether the supposed mechanism of action of this innovative therapy, in relation to the representativity of the endothelial progenitors, carrying the vascular regeneration activity, is preserved in the sclerodermic context.

A total of 30 subjects (20 systemic Scleroderma patients and 10 healthy donors) will be included.

ELIGIBILITY:
Inclusion Criteria:

Patients with systemic scleroderma:

* fulfilling the inclusion criteria for the SCLERADEC 2 trial: patients with systemic Scleroderma older than 18, desiring a therapeutic alternative and having a functional impotence authenticated by a functional index of Cochin's hand greater than 20.
* having given their consent for the constitution of a sample in the biological collection
* having completed the follow-up visit to M3 of the SCLERADEC 2 study to have responder / non-responder status.

Healthy volunteers:

* having recourse to a liposuction operation for aesthetic reasons,
* with a BMI between 18 and 27,
* not declaring chronic diseases,
* having signed the non-opposition

Exclusion Criteria:

Patients with systemic scleroderma:

* Body mass index (weight-to-height ratio squared) less than 18
* Major Sclerodactyly objectified by Rodnan score applied by hand> 16 (out of a total of 18 points)
* Severe tendon retraction of the fingers objectified by a defect extension in passive measure in goniometry> 90 ° C for at least 2 proximal interphalangeal joints
* Digital infection (including infected ulcer, ulcer with local inflammatory signs and clinical suspicion of osteitis)
* Pulmonary arterial hypertension and / or progressive and / or oxygen-dependent pulmonary fibrosis
* Prescription of a new systemic treatment for Systemic Scleroderma in the month prior to inclusion
* Persons infected with HIV, HCV, HBV, HTLV and syphilis
* Patients on immunosuppressants outside corticosteroid therapy <10 mg / day and methotrexate
* Known hypersensitivity to human albumin

For healthy patients and volunteers:

* Contraindication to surgery (patients on anticoagulant or antiaggregant, disorders of haemostasis, contraindication to the analgesic protocol used)
* Premenopausal women of childbearing age without contraception
* Minors
* Pregnant or lactating women
* Majors protected by law (under tutorship or curatorship)
* Persons staying in a health or social facility
* People in emergency
* Persons deprived of their liberty
* Inmates
* Non-beneficiaries of a social security scheme
* Absence or refusal of non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with systemic scleroderma included in the SCLERADEC 2 trial and healthy volunteers who use a liposuction operation for aesthetic reasons.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Study of the gene expression profile | 18 months
  Study of the gene expression profile by qPCR

SECONDARY OUTCOMES:
Phenotypic analysis of the cells composing the stromal vascular fraction | 18 months
  Phenotypic analysis performed by flow cytometry after multiple immunolabelings (CD90, CD14, CD146, CD34, CD45, DRAQ5, NucBlue Fixed Cell Stain (DAPI)) performed in accordance with the recommendations of the International Society for Cellular Therapy (ISCT) and IFATS.
Cell culture of the stromal vascular fraction to isolate and expand two populations of interest | 18 months
  Mesenchymal stem cells (MSCs) obtained by culturing the total stromal vascular fraction without an immunomagnetic selection step.
Cell culture of the stromal vascular fraction to isolate and expand two populations of interest | 18 months
  Endothelial progenitors by a magnetic immuno-separation method (CD144 microbeads kit, Mylteni biotec) for specifically isolating and expanding endothelial progenitor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Direction de la Recherche Clinique et Innovation, Marseille, France